CLINICAL TRIAL: NCT06260267
Title: A Phase 1b Proof-of-concept Trial Exploring the Effects of FE 999322 and FE 999324 in Adults With Mild to Moderate Ulcerative Colitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not due to safety concerns, but changes in strategy which this trial no longer fulfills.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000417
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FE 999322 (Experimental): Microbiota suspension
  Interventions: Drug: Microbiota suspension
- FE 999324 (Experimental): Microbiota capsule
  Interventions: Drug: Microbiota capsule
- Placebo FE 999322 (Placebo Comparator): Placebo suspension
  Interventions: Drug: Placebo suspension
- Placebo FE 999324 (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Microbiota suspension — Microbiota suspension
  Arms: FE 999322
Drug: Microbiota capsule — Microbiota capsule
  Arms: FE 999324
Drug: Placebo suspension — Placebo suspension
  Arms: Placebo FE 999322
Drug: Placebo capsule — Placebo capsule
  Arms: Placebo FE 999324

SUMMARY:
To explore the safety of FE 999322 (microbiota suspension) and FE 999324 (microbiota capsule) versus placebo in subjects with active mild to moderate ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥18 at screening
* Established diagnosis of ulcerative colitis by standard clinical, endoscopic and histological criteria, for more than 3 months at screening

Exclusion Criteria:

* Active disease or history of Crohn's disease
* Active disease or history of irritable bowel syndrome (IBS) or any other chronic intestinal disease apart from UC
* Active gastrointestinal infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events from baseline to week 52 | From baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (10):
- United States (10):
  - Ferring Investigational Site, North Little Rock, Arkansas
  - Ferring Investigational Site, Hamden, Connecticut
  - Ferring Investigational Site, Inverness, Florida
  - Ferring Investigational Site, Jacksonville, Florida
  - Ferring Investigational Site, Orange City, Florida
  - Ferring Investigational Site, Glenview, Illinois
  - Ferring Investigational Site, Gurnee, Illinois
  - Ferring Investigational Site, Shreveport, Louisiana
  - Ferring Investigational Site, Boston, Massachusetts
  - Ferring Investigational Site, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No